CLINICAL TRIAL: NCT04355611
Title: Cohort Study Evaluating the Epidemiological Characteristics of Coronavirus Infection (SARS-CoV-2) in Patients With MS or NMO
Brief Title: Epidemiological Characteristics of COVID-19 in Patients With MS or NMO
Acronym: COVISEP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200482
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis; NMO Spectrum Disorder; COVID-19
Keywords: Factors
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with MS or NMO: Cohort study evaluating the epidemiological characteristics of coronavirus infection (SARS-CoV-2) in patients with MS or NMO
  Interventions: Other: Evaluation of the epidemiological characteristics of coronavirus infection (SARS-CoV-2)

INTERVENTIONS:
Other: Evaluation of the epidemiological characteristics of coronavirus infection (SARS-CoV-2) — Epidemiological characteristics of coronavirus infection (SARS-CoV-2) in patients with MS or NMO

SUMMARY:
The purpose of this study is to collect French medical data for patients with Multiple Sclerosis (MS) or NeuroMyelitis Optica (NMO) spectrum disorder who are diagnosed or strongly suspected of being infected with Covid19. The objective of this study is to provide scientific information regarding the possible risk factors in these patients, as a large part of them receive immunomodulatory or immunosuppressive treatments. The main objective of this study is thus to determine the epidemiological (eg, age, form of disease, disability) and pharmacological (related to immunomodulatory or immunosuppressive treatments) factors favoring the occurrence of a severe form of Covid-19 in MS and NMO patients.

DETAILED DESCRIPTION:
There are currently no data on the consequences of coronavirus infection in patients with Multiple Sclerosis (MS) or NeuroMyelitis Optica (NMO) spectrum disorder. Numerous questions have emerged regarding the management of immunoactive therapy in the case of infection or suspected infection related to the SARS-CoV-2 virus. Currently, the recommendations issued by the French MS Society are to maintain the disease modifying therapies (DMT) for MS and NMO, but a case-by-case discussion with the expert neurologist for suspected or confirmed COVID+ patients remain highly recommended. Besides DMT, neurological disability could also be a risk factor for severe infection, regardless of the age of the patient.

It is therefore essential to have epidemiological data to describe the characteristics of the clinical expression of coronavirus infection (Covid-19) and factors enhancing the occurrence of severe forms in patients with MS or NMO during of the 2020 pandemic.

This study involves all hospital and neurologists ensuring the follow-up of patients with MS and NMO via the 23 CRC-SEP and associated hospital centers. This multicenter study is based on an already functional network organization, grouping together around forty hospital centers, participating either in the French MS registry (OFSEP), or in the French MS Society (SFSEP). It also benefits from the support of the French clinical research network (FCRIN) through the thematic clinical research network on MS and related diseases (FCRIN4MS). Each day, participating centers will enter data from MS or NMO patients newly tested positive for SARS-CoV-2 or strongly suspected to be diagnosed with COVID-19 using a specific computerized record (CRF Redcap).

ELIGIBILITY:
Inclusion criteria

* Patient with MS or NMO
* at least one of the following four criteria:

  * COVID + biologically confirmed
  * Typical ground glass opacity on thoracic CT-scan in epidemic areas
  * Anosmia or ageusia of sudden onset in the absence of rhinitis or nasal obstruction
  * Typical symptoms (triad associating cough, fever, asthenia) in epidemic zone
* Non opposition of the patient to the use of these data or non opposition of the confidential counselor / parent / relative (if the patient is unable to give his non-opposition, with collection as soon as possible of the non opposition of the patient) or non opposition of the 2 holders of parental authority (for minor patients)

Non-inclusion criteria

- Patient under guardianship or safety measure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Multiple Sclerosis (MS) or NeuroMyelitis Optica (NMO) spectrum disorder who are diagnosed or strongly suspected of being infected with Covid19.
Sampling Method: Non-Probability Sample
Enrollment: 2465 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical severity | 6 months
  The main outcome measure is a clinical severity score on a 7-point severity scale at Nadir (in medicine, the most severe point in the progression of symptoms of a pathology).
  Nadir scale from 1 : Not hospitalized, no limitation of activities to 7 :Death

SECONDARY OUTCOMES:
EDSS (Expanded Disability Status Scale) | 6 months
  EDSS is the Expanded Disability Severity Scale, a measure of neurological disability in patients with MS or NMO.
  EDSS Scale from 0: normal neurological examination to 10: MS-related Death

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié Salpétrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided